CLINICAL TRIAL: NCT03518697
Title: Effects of an Individualized and Partially Supervised Exercise Program on Parameters of Physical Fitness, Lung Function, Habitual Physical Activity in Daily Life and Quality of Life in Children, Adolescents and Adults With Cystic Fibrosis.
Brief Title: Effects of an Individualized Exercise Program on Health-related and Skill/Performance-related ﬁtness in CF.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Essen (Other)
Responsible Party: Principal Investigator, Florian Stehling, Dr. Florian Stehling, Head of Pediatric Pulmonology, Children´s Hospital, University Hospital, Essen
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 14-6117-BO
Record Dates: First submitted 2018-03-26; First posted 2018-05-08 (Actual); Last update posted 2019-01-03 (Actual); Status verified 2019-01

CONDITIONS: Cystic Fibrosis
Keywords: Exercise; Physical fitness; Physical activity; Accelerometer; Sleep
MeSH Terms: conditions — Cystic Fibrosis; Motor Activity | interventions — Resistance Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise Group (Experimental): 1. First 6 months supervised exercise program with telephone contact every two weeks
  2. Second 6 months exercise program without telephone contact
  3. Patients should increase habitual daily physical activity for 10-20 minutes per day 5 times per week
  4. Activities were chosen according to the preferences, interests, and severity of disease of the patients
  5. Activites should improve endurance, strength, coordination and flexibility
  6. Every three month regular vistit at the CF care center (medical examination, lung function, exercise testing, counselling and evaluation of activities by acceleometry and if appropirate adaption of exercise program)
  Interventions: Behavioral: exercise program
- Control-Group (No Intervention): 1. 12 months usual routine care and habitual exercise in daily life.
  2. At start and after 12 month assessment of habitual exercise with accelerometry (Actigraph GTX3)

INTERVENTIONS:
Behavioral: exercise program — The exercise program is planned as a "low-threshold exercise program "with low barriers to participate. Patients will be asked about their interests and preferences of sports activities to conceive the exercise program together with the patients.
  Arms: Exercise Group

SUMMARY:
The aim of this study is to evaluate the effects of a partially supervised exercise program on different aspects of physical fitness, despite VO2peak, lung function, quality of life and sleep quality in children, adolescents and adults with Cystic Fibrosis.

DETAILED DESCRIPTION:
There is growing consensus that exercise in subjects with cystic fibrosis (CF) may yield improvements in measures of physical fitness, lung function and quality of life. In most of the training studies exercise capacity was expressed as peak oxygen uptake (VO2peak), which has been found to be one of the best predictors of survival in subjects with CF. Those subjects with a higher VO2peak related to age and gender specific predicted VO2peak (%pred) have a better prognosis than those with a lower VO2peak (%pred). VO2peak represents the cardiorespiratory endurance is one aspect of physical fitness.

Physical ﬁtness may be subdivided into health-related ﬁtness and skill/performance-related ﬁtness. Cardiorespiratory endurance, muscular strength and endurance, body composition and ﬂexibility are often referred to as health-related ﬁtness. Balance, coordination, speed, agility and power are often described as skill/performance related ﬁtness, reﬂecting the performance aspect of physical ﬁtness. It has been shown, that children and adolescents with a lower skill / performance related fitness are less physical active than those with a higher skill/performance related fitness. This may lead to physically inactive in daily life, less motivation to take part in organized sport and as a consequence to a lower VO2peak.

The primary outcome parameters of this study is to evaluate the effects 12-month partially supervised exercise program on 1) health-related ﬁtness (endurance expressed as maximal workload, muscular strength) and skill / performance related fitness (balance, power, agility)and 2) habitual physical activity (steps / day; intensity expressed in METs) in a large group of subjects with CF. Secondary outcome parameters include forced exspiratory volume in 1 second (FEV1), sleep-wake cycle, quality of sleep, quality of life, and exercise related barriers and barrier management in physical exercise.

In total 100 subjects with CF 6 year and older will be included. Habitual physical activity and sleep will be recorded by accelerometer before subjects enter the exercise program, and after 6 month and after 12 month. Check-ups, lung function measurement and testing of physical fitness will be performed at baseline, after 6 and 12 month.

During the first six month the participants will be contacted by telephone every two weeks. After six month individual counseling by telephone will be stopped.

The exercise program is planned as a "low-threshold exercise program "with low barriers to participate. Participants will be asked about their interests and preferences of sports activities to conceive the exercise program together with the participants. Along with counseling participants will be motivated to increase physical activity by at least 10-20 minutes per day.

The investigators expect to gain another insight into different aspects of physical fitness, habitual physical activity and sleep from the results of this study. Up to know, there are only a few trails investigated different aspects of physical fitness that means balance, flexibility, power as parameters of health-related ﬁtness and skill/performance-related ﬁtness. The investigators assume that participants with higher values are more physical active than those with lower values and these participants will have a higher cardiorespiratory endurance.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of CF
* Informed consent

Exclusion Criteria:

* Cardiac arrhythmias with exercise
* Patients with cor pulmonale
* Colonization with Burkholderia cenocepacia, Methicillin-resistant Staphylococcus aureus (MRSA) and multidrug-resistant Gram-negative (MRGN) pathogens (3 and 4 MRGN)
* Patients with untreated diabetes

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2014-09-10 (Actual); Primary Completion 2018-08-10 (Actual); Study Completion 2018-08-10 (Actual)

PRIMARY OUTCOMES:
Change of habitual physical activity in hours/day | at baseline, after 6 and 12 month
  Measurement of the time of physical activity in hours/day by accelerometry (ActiGraph GT3X, Penascola, USA)

SECONDARY OUTCOMES:
Change of the quality of life in Cystic Fibrosis | at baseline, after 6 and 12 month
  Measurement of the quality of life by the Cystic Fibrosis Questionnaire Revised (CFQ-R, Quality of life domains: Physical, role/school, vitality, emotion, social, body image, eating, treatment burden, health perceptions. Symptom scales: Weight, respiratory, and digestion)
Change of the duration of sleep in hours | at baseline, after 6 and 12 month
  Measurement of the duration of sleep in hours by accelerometry (ActiGraph GT3X, Penascola, USA)
Change of the quality of sleep in percent | at baseline, after 6 and 12 month
  Measurement of the quality of sleep in percent by accelerometry (ActiGraph GT3X, Penascola, USA)
Determination of the exercise related barriers and barrier management in physical exercise | at baseline
  specific questionnaire (Barrieren und Barrierenmanagementim Prozess der Sportteilnahme, Krämer and Fuchs, Zeitschrift für Gesundheitspsychologie, 18(4), 170-182, 2010)
Change of habitual physical activity in steps/day | at baseline, after 6 and 12 month
  Measurement of the number of steps/day by accelerometry (ActiGraph GT3X, Penascola, USA)
Change of habitual physical activity spend in light intensity (≤ 3METS) in minutes | at baseline, after 6 and 12 month
  Measurement of the time of habitual physical activity spend in light intensity (≤ 3METS) in minutes by accelerometry (ActiGraph GT3X, Penascola, USA)
Change of habitual physical activity spend in moderate to vigorous intensity (3 to 5.9 METS) in minutes by accelerometry (ActiGraph GT3X, Penascola, USA) | at baseline, after 6 and 12 month
  Measurement of the time of habitual physical activity spend in moderate to vigorous intensity (3 to 5.9 METS) in minutes by accelerometry (ActiGraph GT3X, Penascola, USA)
Change of habitual physical activity spend in vigorous intensity (6 to 8.99 METS) in minutes by accelerometry (ActiGraph GT3X, Penascola, USA) | at baseline, after 6 and 12 month
  Measurement of the time of habitual physical activity spend in vigorous intensity (6 to 8.99 METS) in minutes by accelerometry (ActiGraph GT3X, Penascola, USA)
Change of habitual physical activity spend in hard intensity (≥ 9 METS) in minutes by accelerometry (ActiGraph GT3X, Penascola, USA) | at baseline, after 6 and 12 month
  Measurement of the time of habitual physical activity spend in hard intensity (≥ 9 METS) in minutes by accelerometry (ActiGraph GT3X, Penascola, USA)
Change of maximal exercise capacity expressed as heart rate | at baseline, after 6 and 12 month
  Measurement of heart rate in b/min by cycle ergometry (Ergoselect 100p, Ergoline, Bitz, Germany)
Change of maximal exercise capacity expressed as heart rate reserve in percent | at baseline, after 6 and 12 month
  Measurement of heart rate reserve in percent by cycle ergometry (Ergoselect 100p, Ergoline, Bitz, Germany)
Change of maximal exercise capacity expressed as workload in Watt | at baseline, after 6 and 12 month
  Measurement of workload in Watt by cycle ergometry (Ergoselect 100p, Ergoline, Bitz, Germany)
Change of maximal exercise capacity expressed as workload in Watt / kg bodyweight | at baseline, after 6 and 12 month
  Measurement of workload in Watt / kg bodyweight by cycle ergometry (Ergoselect 100p, Ergoline, Bitz, Germany)
Change of maximal exercise capacity expressed as perceived exertion (Borg CR10 Scale) in number of level of exertion | at baseline, after 6 and 12 month
  Measurement of the Borg questionnaire (Borg CR10 Scale)
Change of skill / performance related fitness expressed as push-ups in number of repetition in 40 sec. | at baseline, after 6 and 12 month
  Measurement of push-ups in number of repetition in 40 sec. with the German motor test (Deutscher Motorik Test, Forschungszentrum für den Schulsport und den Sport von Kindern und Jugendlichen, Karlsruhe, Germany) in children and adolescents aged 6-18 years
Change of skill / performance related fitness expressed as standing broad jump in cm in children and adolescents | at baseline, after 6 and 12 month
  Measurement of standing broad jump in cm with the German motor test (Deutscher Motorik Test, Forschungszentrum für den Schulsport und den Sport von Kindern und Jugendlichen, Karlsruhe, Germany) aged 6-18 years
Change of skill / performance related fitness expressed as sit-up in number of repetition in 40 sec. | at baseline, after 6 and 12 month
  Measurement of sit-ups in number of repetition in 40 sec. with the German motor test (Deutscher Motorik Test, Forschungszentrum für den Schulsport und den Sport von Kindern und Jugendlichen, Karlsruhe, Germany) aged 6-18 years
Change of skill / performance related fitness expressed as balancing backwards number in steps on a wooden beam 6 cm wide and 3 meters long | at baseline, after 6 and 12 month
  Measurement of balancing backwards number in steps on a wooden beam 6 cm wide and 3 meters long with the German motor test (Deutscher Motorik Test, Forschungszentrum für den Schulsport und den Sport von Kindern und Jugendlichen, Karlsruhe, Germany) aged 6-18 years
Change of skill / performance related fitness expressed as jump sideways in number of repetition in 15 sec. | at baseline, after 6 and 12 month
  Measurement of balancing backwards number in jump sideways in number of repetition in 15 sec. with the German motor test (Deutscher Motorik Test, Forschungszentrum für den Schulsport und den Sport von Kindern und Jugendlichen, Karlsruhe, Germany) aged 6-18 years
Change of skill / performance related fitness expressed as flexibility in cm in children and adolescents | at baseline, after 6 and 12 month
  Measurement of flexibility in cm with the German motor test (Deutscher Motorik Test, Forschungszentrum für den Schulsport und den Sport von Kindern und Jugendlichen, Karlsruhe, Germany) aged 6-18 years
Change of skill / performance related fitness expressed as one leg stand in sec. | at baseline, after 6 and 12 month
  Measurement of one leg stand in sec. as included in the TFR (Test Fitness Rekrutierung, Bundesamt für Sport BASPO, Magglingen, Schweiz) in adults
Change of skill / performance related fitness expressed as standing broad jump in cm in adults | at baseline, after 6 and 12 month
  Measurement of standing broad jump in cm as included in the TFR (Test Fitness Rekrutierung, Bundesamt für Sport BASPO, Magglingen, Schweiz) in adults
Change of skill / performance related fitness expressed as trunk power in sec. | at baseline, after 6 and 12 month
  Measurement of trunk power in sec. as included in the TFR (Test Fitness Rekrutierung, Bundesamt für Sport BASPO, Magglingen, Schweiz) in adults
Change of skill / performance related fitness expressed as flexibility in cm in adults | at baseline, after 6 and 12 month
  Measurement of flexibility in cm as included in the basic motor diagnostics (Motorische Basisdiagnostik, Hrsg. Bös/Wydra/Karisch, 1992) in adults
Change of skill / performance related fitness expressed as circling motion in number of complete performed circles | at baseline, after 6 and 12 month
  Measurement of circling motion in number of complete performed circles as included in the basic motor diagnostics (Motorische Basisdiagnostik, Hrsg. Bös/Wydra/Karisch, 1992) in adults
Change of skill / performance related fitness expressed as the time of hip extension in sec. | at baseline, after 6 and 12 month
  Measurement of the time of hip extension in sec. as included in the basic motor diagnostics (Motorische Basisdiagnostik, Hrsg. Bös/Wydra/Karisch, 1992) in adults

CONTACTS AND LOCATIONS:
Locations (3):
- Germany (3):
  - St. Josef-Hospital im Katholischen Klinikum Bochum, Klinik für Kinder und Jugendmedizin, Alexandrinenstrasse 5, Bochum
  - Universitätsklinikum Essen, Klinik für Kinderheilkunde III, Pädiatrische Pneumologie und Schlafmedizin, Hufelandstr. 55, Essen
  - Ruhrlandklinik Essen, Westdeutsches Lungenzentrum am Universitätsklinikum Essen, Tuschener Weg 40, Essen

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dietz-Terjung S, Gruber W, Sutharsan S, Taube C, Olivier M, Mellies U, Koerner-Rettberg C, Dillenhofer S, Stehling F, Welsner M. Association between habitual physical activity (HPA) and sleep quality in patients with cystic fibrosis. Sleep Breath. 2021 Jun;25(2):609-615. doi: 10.1007/s11325-020-02130-0. Epub 2020 Jul 14. PMID 32661789